CLINICAL TRIAL: NCT02584179
Title: Can Significant Prostate Cancer be Detected With a Short Non-contrast Enhanced Biparametric MRI (bpMRI)?
Brief Title: Biparametric MRI for Detection of Significant Prostate Cancer
Acronym: BIDOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Karen-Cecilie Duus Thestrup, Cand. med., Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Herlev-MR-Prost-BP
Record Dates: First submitted 2015-09-06; First posted 2015-10-22 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: mpMRI, significant cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biparametric MRI before biopsy (Experimental): Biparametric MRI is a reduced Multiparametric MRI using less scan sequences and no intravenous contrast.
  All men will have standard transrectal ultrasound guided biopsies
  Interventions: Device: Biparametric MRI before biopsy

INTERVENTIONS:
Device: Biparametric MRI before biopsy — All included men with suspicious lesions on bpMRI will have bpMRI targeted biopsies in addition to standard TRUS-bx.
  Other Names: BpMRI

SUMMARY:
Our aim is to develop a new diagnostic approach to improve the diagnosis of men suspicious of having significant prostate cancer (sPCa). The current diagnostic technique (standard transrectal ultrasound-guided biopsies [TRUS-bx]) rely on multiple prostate biopsy cores (10-12 samples) and if negative repeated biopsy sessions. This increases both patient complications (severe infections, bleeding and anxiety) and the diagnosis of insignificant cancer causing overtreatment. Still, significant cancers are missed. In addition, worldwide antibiotic-resistant bacteria increase, while effective antibiotics are declining. Thus, a noninvasive diagnostic tool to improve selection of men with clinically suspicion of PCa who need a biopsy from those who can avoid one is strongly needed. Previous studies in our department show that MRI in a selected patient cohort with prior negative TRUS-bx can improve the detection rate of clinically significant PCa and allows for a more accurate assessment of cancer stage and aggressiveness. However, the value of an MRI used as a first-line tool in the diagnostic examination of men in suspicion of PCa is uncertain. Furthermore, a full scale MRI prostate examination recommended by the European Society of Urogenital Radiology includes intravenous contrast-media and multiple sequences. This is both time-consuming and cost full, which reduces its feasibility for more widespread clinical implementation. We believe that a simpler, faster biparametric MRI (bpMRI) using less scan sequences and circumvents intravenous contrast-media and anti-peristaltic drugs would decrease image acquisition time, reduce costs and is sufficient to preserve diagnostic accuracy for sPCa detection in biopsy-naive men. Consequently, we will include biopsy-naive men in a protocol-based research project. The objective is to assess the diagnostic accuracy of bpMRI to rule out sPCa and whether a bpMRI can be used as a diagnostic non-invasive screening tool to 1) improve the diagnosis of sPCa 2) assess cancer aggressiveness 3) increase precision of biopsies and 4) reduce the number of biopsy sessions and cores. We evaluate the clinical significance of the detected cancers and whether bpMRI could be used as a triage test to improve the diagnosis of sPCa and aid in the determination of which men could safely avoid unnecessary biopsies.

This new diagnostic approach has the potential to significantly reduce patient hazards and complications. We aim to reach 1000 included men. We believe that bpMRI used in the clinical decision-making has the potential to change the future management of PCa. However, we still miss the scientific evidence to substantiate its preliminary promising results before this technique can be widely used to benefit all men. This large research project is to the best of our knowledge powered to include the largest patient sample size published within this field.

DETAILED DESCRIPTION:
Purpose Our aim is to assess whether a screening bpMRI can be used as a diagnostic non-invasive screening tool to 1) improve the diagnosis of sPCa 2) predict cancer aggressiveness 3) increase precision of biopsies and 4) reduce the number of biopsy sessions and cores.

Trial subjects Subjects are recruited at the Department of Urology, Herlev Gentofte University Hospital. Annually, approx. 1.600 men are referred to the department due to clinical suspicion of PCa. Roughly 1.100 men further proceeds to standard TRUS-bx prostate biopsies. These men are invited to participate as subjects in this study and undergo a bpMRI before biopsies, if they fulfil the inclusion criteria. All subjects provide written informed consent and can withdraw their consent at any time with no consequence in relation to their standard treatment. Intended sample size calculations (power 0•9 and 2-sided significance 0•05) were based on estimates of diagnostic accuracy (sensitivity and specificity) and detection rates by biopsy techniques (SBx and TBx) from prior mpMRI studies assuming prevalence of sPCa of 30%. Target sample size was minimum 600 patient.

Study Design This study is designed as a prospective interventional study. All enrolled patients undergo a screening bpMRI of the prostate within 1-2 weeks after inclusion and prior to biopsies. All MRI data undergo blinded evaluation according to a modified PIRADS version 2 classification from the European Society of Urogenital Radiology (ESUR) 18 by an experienced physician who register and score all suspicious lesions on a five-point scale (1- very low, 2 - low, 3 - intermediate, 4- high and 5 - very high) according to the overall probability of having significant PCa. As the bpMRI protocol does not include dynamic contrast-enhanced (DCE) imaging, scoring of lesions in the peripheral zone relied solely on DWI findings. The bpMRI is within 4-weeks followed by standard 10-core TRUS-bx performed according to current standard practice and blinded to any MRI findings. The TRUS-operator then subsequently reviews the MRI data and rapport on a dedicated workstation in the biopsy room to identify suspicious lesions presented and outlined by the radiologist. Any suspicious lesions are then targeted by additional bpMRI-guided biopsies using bpMRI-TRUS image fusion based software. BpMRI suspicion scores and biopsy results from TRUS-bx and bpMRI-bx are compared.

Furthermore, all enrolled patients are clinically followed for 5 years after the initial biopsies to detect any subsequent diagnosis of PCa, treatment recurrence or metastasis.

MRI image acquisition:

A 3T MRI-scanner (Ingenia, Philips Healthcare, the Best, the Netherlands) is used for all patients with a pelvic-phased-array coil (Philips Healthcare, Best, the Netherlands) positioned over the pelvis. Anatomical (T2W) and diffusion-weighted images (DWI) including 4 b-values (b0, b100, b800 and b2000) along with reconstruction of the corresponding apparent diffusion coefficient (ADC) map (b-values 100 and 800) are obtained from below the prostatic apex to above the seminal vesicles. A sagittal T2W luxury scout supported the axial sequences for MRI/TRUS image fusion.

Pathological evaluation A genitourinary pathologist with more than 11 yrs of dedicated experience in prostatic pathology reviews and describes all histological biopsy samples. For each PCa positive biopsy core, the location and prostatic region, the Gleason score (GS) 19 and the extent of cancer core involvement (%) are determined. Various definitions of sPCa are assessed including GS and tumor volume.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 85 years.
* Clinical suspicion of PCa based on: serum level of prostate-specific-antigen (PSA) from 2.5 ng/ml in two consecutive measurements and/or abnormal diagital rectal examination (DRE).
* Mental status: Patients must be able to understand the objective of the study.
* Informed consent: The patient must sign the local Ethics Committee (EC) approved informed consent documents in the presence of the designated staff.

Exclusion Criteria:

* Previous prostate biopsies.
* Previous diagnosis of PCa.
* Acute prostatitis.
* Contraindications to MRI (cardiac pacemaker, claustrophobia etc).
* Infection (temperature > 38 degrees Celsius)
* Hip replacement surgery or other metal implants in the pelvic area.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1063 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of a bp-MRI in detection and ruling out significant PCa in biopsy-naive men | 24 months
  All included men undergo bp-MRI at inclusion followed by diagnostic standard TRUS biopsies (current diagnostic standard). Men with any suspicious lesions on bpMRI undergo additional bpMRI-guided biopsies (bpMRI-bx) using bpMRI-TRUS image fusion based software. BpMRI suspicion scores and biopsy results ( detection of any PCa and sPCa) from standard TRUS-bx and bpMRI-bx are compared using combined biopsy results as standard reference.
  Sensitivity and negative predictive value of bpMRI to detect and rule out sPCa will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Thomsen, MD, Study Chair — Herlev Hospital, Herlev Ringvej 75, 2730 Herlev, Denmark; Lars Boesen, MD, PhD, Study Chair — Deptartment of Urology, Herlev Hospital, Herlev Ringvej 75, 2730 Herlev, Denmark
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
as a publication